CLINICAL TRIAL: NCT07146971
Title: Clinical Evaluation of the Skin Microbiome and the Efficacy of an Over-The-Counter (OTC) Drug for Atopic Dermatitis
Brief Title: Clinical Evaluation of Skin Microbiome an Over-The-Counter (OTC) Drug for Atopic Dermatitis
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Good Molecules, LLC (Industry)
Collaborators: Sequential Skin Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SS-NLP-417
Record Dates: First submitted 2025-08-15; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Atopic Dermatitis (AD)
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Nonprescription Drugs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Atopic Dermatitis OTC Product (Experimental)
  Interventions: Drug: OTC Drug for Atopic Dermatitis in Cream form
- No Product (No Intervention)

INTERVENTIONS:
Drug: OTC Drug for Atopic Dermatitis in Cream form — OTC Cosmetic Cream Formulation
  Arms: Atopic Dermatitis OTC Product

SUMMARY:
This is a research study. The over-the-counter (OTC) drug for atopic dermatitis being tested is not approved as a treatment for the participants' atopic dermatitis condition. In participating in this study, the investigators will analyze the participants' skin microbiome, measure skin hydration and barrier function, and assess clinical improvements to help us understand the potential impact of the investigational OTC drug on atopic dermatitis and skin microbiome balance.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed Atopic Dermatitis with active, visible flare-ups at time of screening
* Present dry/itchy skin patches on forearms suitable for treatment assessment
* Evidence of inflammatory disease (documented diagnosis and current active symptoms)
* Stable skincare routine for 4 weeks prior to screening
* Subject willing to avoid conflicting topical treatments during study period
* Subject being used to applying topical treatments for atopic dermatitis

General:

* Healthy subject apart from atopic dermatitis
* Subject having given free informed, written consent
* Subject willing to adhere to protocol and study procedures

Exclusion Criteria:

* Pregnant or nursing woman or woman planning to get pregnant during the study
* Recent (within 4 weeks) or current history of using atopic dermatitis biological drugs, such as dupilumab, lebrikizumab, nemolizumab, and tralokinumab
* Recent use of systemic antibiotics, steroids, or immunomodulators (within 4 weeks)
* Active skin infections unrelated to atopic dermatitis
* Severe dermatologic conditions requiring immediate medical intervention
* Use of topical or systemic treatment during previous weeks liable to interfere with assessment
* Subject having undergone surgery under general anaesthesia within the previous month
* Excessive exposure to sunlight or UV-rays within the previous month
* Subject having scars, tattoos on the forearms that would interfere with assessments
* Subject enrolled in another clinical trial during the study period and/or during the past 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-28 (Estimated); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-11-25 (Estimated)

PRIMARY OUTCOMES:
Skin Microbiome Composition and Diversity using qPCR analysis | 4 weeks
Trans-Epidermal Water Loss Measurement via Vapometer | 4 weeks
Moisturizing effect by measurement of cutaneous hydration via MoistureMeterSC | 4 weeks
Skin barrier lipid composition and integrity via lipidomic profiling analysis | 4 weeks

SECONDARY OUTCOMES:
Before and After Treated Arm Itching Assessment | 4 weeks
  In vivo clinical grading by a technician using a 11 point scale (0 = uncomfortable, irritated, and 10 = comfortable, soothed)
Before and After Treated Arm Redness Assessment | 4 weeks
  In vivo clinical grading by a technician using a 5 point scale (0 = absence of redness, and 4 = severe intensity)
Before and After Treated Arm Skin Dryness Assessment | 4 weeks
  In vivo clinical grading by a technician using a 11 point scale (0 = dry, cracked skin, and 10 = well-hydrated skin)
Monitoring of Atopic Dermatitis/Eczema Severity | 4 weeks
  Via the Patient Oriented Eczema Measure (POEM) tool

CONTACTS AND LOCATIONS:
Locations (1):
- Sequential Skin, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT07146971/ICF_000.pdf